CLINICAL TRIAL: NCT07175987
Title: A Consumer Use Behavior Study to Evaluate Puffing Topography and Average Daily Consumption of Heated Tobacco Products in the UK
Brief Title: A Consumer Use Behavior Study to Evaluate Puffing Topography and Average Daily Consumption of Heated Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: IPSOS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHCB2IT20257
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cigarette
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HTP Device (1) (Experimental): Participants will be randomized to one of three stick variants.
  Interventions: Other: RDTH002581; Other: RDTH002580; Other: RDTH002582
- HTP Device (2) (Experimental): Participants will be randomized to one of three stick variants.
  Interventions: Other: RDTH002578; Other: RDTH002577; Other: RDTH002579

INTERVENTIONS:
Other: RDTH002581 — Participants assigned to this Study Intervention will use the product only in the CLT portion of the study.
  Arms: HTP Device (1)
Other: RDTH002580 — Participants assigned to this Study Intervention will use the product in the CLT and HUT portions of the study.
  Arms: HTP Device (1)
Other: RDTH002582 — Participants assigned to this Study Intervention will use the product in the CLT and HUT portions of the study.
  Arms: HTP Device (1)
Other: RDTH002578 — Participants assigned to this Study Intervention will use the product only in the CLT portion of the study.
  Arms: HTP Device (2)
Other: RDTH002577 — Participants assigned to this Study Intervention will use the product in the CLT and HUT portions of the study.
  Arms: HTP Device (2)
Other: RDTH002579 — Participants assigned to this Study Intervention will use the product in the CLT and HUT portions of the study.
  Arms: HTP Device (2)

SUMMARY:
This is a parallel design cohort consumer use study to measure the puffing topography of two HTP devices, with three variants of HTP consumables ("sticks,"), collectively referred to as the study investigational products (Study IP), among a sample of n=198 primary users of combustible cigarettes at a central location testing (CLT) facility in the United Kingdom (UK). Puffing topography at the CLT will be measured using a desktop puffing analyzer device (PA1).

In addition to puffing topography measurements at the CLT, a tobacco product perceptions and intentions survey will be used to assess study participants' intent to purchase the Study IP, their risk perceptions, and their intended use behaviors. Participants' demographic characteristics (including age and biological sex), and tobacco- and nicotine-containing products (TNPs) use history will be collected using self-reported questionnaires.

Following completion of the CLT, a subset (n=100) of the originally enrolled population will participate in a 5-day home use testing (HUT) period in which they will use the Study IP for 5 days in their everyday environments to assess average daily consumption (ADC) and usage patterns of the Study IP, as well as use of any other TNPs, recorded in a daily survey. On completion of the last day of the HUT, participants will complete a final end of study survey assessing product liking, purchase intent, and intended use behaviors.

DETAILED DESCRIPTION:
This is a parallel design cohort consumer use study to measure the puffing topography of two HTP devices (glo and glo plus), with three variants of HTP consumables ("sticks," under the brand name "virto"), collectively referred to as the study investigational products (Study IP), among a sample of n=198 primary users of combustible cigarettes at a central location testing (CLT) facility in the United Kingdom (UK). Puffing topography at the CLT will be measured using a desktop puffing analyzer device (PA1).

In addition to puffing topography measurements at the CLT, a tobacco product perceptions and intentions survey will be used to assess study participants' intent to purchase the Study IP, their risk perceptions, and their intended use behaviors. Participants' demographic characteristics (including age and biological sex), and tobacco- and nicotine-containing products (TNPs) use history will be collected using self-reported questionnaires.

Following completion of the CLT, a subset (n=100) of the originally enrolled population will participate in a 5-day home use testing (HUT) period in which they will use the Study IP for 5 days in their everyday environments to assess average daily consumption (ADC) and usage patterns of the Study IP, as well as use of any other TNPs, recorded in a daily survey. On completion of the last day of the HUT, participants will complete a final end of study survey assessing product liking, purchase intent, and intended use behaviors.

To account for respondent drop-out, the fieldwork team will recruit approximately 15% more participants for the CLT and approximately 20% more participants to the HUT phase.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 21-65 years (inclusive)
* Be self-reported current 'daily users' of at least 5 CPD and have smoked at least 100 cigarettes in their lifetime. ('daily users' defined as have smoked 5 CPD for at least 27 days out of last 30 days)
* Agree to participate in the study and to abide by the study restrictions and requirements, including the use of the assigned Study IP, as described in the ICF.
* Agree not to allow any other person to use any product provided to them for use during this study.

Exclusion Criteria:

* Women who self-report they are pregnant or breastfeeding or could become pregnant or start breastfeeding in the next three months from the study start date.
* Women who self-report they are not using adequate methods to prevent pregnancy, which they intend to continue throughout the study.

  a. Examples of acceptable means of birth control are, but not limited to: i. Surgical sterilization (hysterectomy, bilateral tubal litigation/occlusion, bilateral oophorectomy, bilateral salpingectomy); ii. Established use of oral, implantable, injectable, or transdermal methods of contraception associated with inhibition of ovulation; iii. Physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide; iv. Non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena); v. Vasectomized partner; vi. Abstinence from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation; and vii. Post-menopausal and not on hormone replacement Therapy
* People who self- report having pacemakers or other embedded electronic medical devices.
* People who self-report having heart disease, high blood pressure, diabetes, depression, or asthma.
* People who have ever used HTP.
* People who self-report currently quitting or planning to quit all nicotine products in the next 3 months.
* People who self-report having participated in tobacco product research in the past 3 months.
* People who self-report themselves, or someone in their direct family or close friends, as working in one of the following areas:

  1. Advertising
  2. Journalism
  3. Media
  4. Insurance
  5. Marketing
  6. Market Research
  7. Manufacturer or retailer of tobacco or vapor products
  8. Public Relations
  9. Sale of Alcohol

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
To measure the puffing topography of primary combustible cigarette smokers when using either of the investigational HTP devices with one of three stick variants during CLT. | 90 minutes
  The primary endpoints will be measured in CLT using a desktop PA1. The data will be summarized using the overall mean per study arm (Study IP device) as well as mean per stick variant within arms.

SECONDARY OUTCOMES:
To determine the average daily consumption of sticks during HUT. | 5 days
  Participants will be asked to log the number of sticks used during the 5-day home use testing period.
To assess purchase intent for participants using each of the study products before and after using the products. | Through study completion
  Participants will be asked before and after using the product how likely they are to purchase the product on a scale from 1 to 10.
To describe subjective characteristics associated with product use, including overall liking | At study completion
  Participants will be asked their overall liking of the product on a 1-10 scale.
To assess risk perceptions before using the products only. | Baseline
  Utilization of Tobacco Product Perception and Intentions (TPPI) survey data to understand the likelihood of certain tobacco and nicotine related use behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Tapia, Ph.D., Study Director — RAI Services Company
Locations (1):
- Channing Hall, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No